CLINICAL TRIAL: NCT05068050
Title: Clinical, Data Collection, Multicenter, Randomized Trial to Determine the Effect of Therapeutic Riding Compared With Physical Activity on a Group of People With Arthritis
Brief Title: Multicenter, Randomized Trial to Determine the Effect of Therapeutic Riding, on a Group of People With Arthritis
Acronym: ARTHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Collaborators: University of Évora (Other); University of Oviedo (Other); AINISE - Alianza Internacional por la Interacción Saludable con Equinos (Unknown); Universidad Rey Juan Carlos (Other); University of Burgos (Unknown); National University of Rosario (Unknown)
Responsible Party: Principal Investigator, Mª Dolores Apolo Arenas, Principal Investigator, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UdeExtremadura-2021-1
Record Dates: First submitted 2021-09-15; First posted 2021-10-05 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Arthritis
Keywords: Therapeutic riding; Horse-assisted therapy; Arthritis treatments; Therapeutic exercise; Inertial Measurement Unit; Gait analysis; Sleep analysis; Pain analysis; Joints analysis
MeSH Terms: conditions — Arthritis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Two groups of participants: i) experimental group, ii) active control group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants do not know the direction of the hypotheses
  The assessors are blinded to the assignment of the participants to the experimental group or the control group.
  The investigators treating the data are blinded to the allocation of participants to the experimental group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This arm will be provided by horse-assisted therapy interventions.
  Interventions: Procedure: Horse-assisted therapy
- Control group (Active Comparator): This arm will be provided by the physical exercise interventions.
  Interventions: Procedure: Physical exercise

INTERVENTIONS:
Procedure: Horse-assisted therapy — 12 horse-assisted therapy sessions (45 mins each) for 6 weeks.
  Each session will comprise the next stages:
  Groundwork, Approachment and preparation of the horse, Warm up exercises
  Development of the main part (riding):
  Introduction - beginning: Breathing control and body awareness, maintain sitting (riding position) while walking on the horse, perceiving the movement Exercises for the postural and balance control: Variations in the walking of the horse, realize different figures in the arena (circles, serpentines, change direction…), Stopping and Walking, Arms situation combined with the movement of the horse All exercises are determined in the track design protocol Exercises for the acquisition of motion skills: Finished the riding with relaxation activities. Final part: Dismount the horse, Unsaddled and unbridle, feedback and goodbye procedure.
  Arms: Experimental group
Procedure: Physical exercise — 12 physical exercise sessions (45 mins each) for 6 weeks. Each session Each session Lessons will be held by physical activity professionals. The proposed exercises are focussed on improving the articular movements, aerobic resistance and the proprioception, always on the premises of No Pain.
  Lessons will be divided in three parts :
  1. Warmup - 2. Main part - 3. Return to calm
  Lessons will be hold online
  Arms: Control group

SUMMARY:
The aim of this job is to evaluate the possible changes in the state of health of 10 indi-viduals diagnosed with arthritis who follow a standardised Therapeutic Riding treatment, as an experimental group, versus 10 patients who follow a standardised physical exercise programme.

The intervention guidelines for both groups are established in a programme of 12 ses-sions in total, 6 weeks in duration, twice a week and a duration of 45 minutes each ses-sion.

The effectiveness of the intervention program will be evaluated in terms of pain, joint mobility, static and dynamic balance, gait, capacity for effort and quality of sleep.

DETAILED DESCRIPTION:
Arthritis is inflammation of the joints, causing pain, stiffness and limitations in activities of daily living, with decreased quality of life.

To improve musculoskeletal and functional health, the World Health Organization recommends physical activity, including aerobic physical activity, to improve strength, flexibility and balance. Non-pharmacological recommendations include physical conditioning, which can be provided through Therapeutic Riding. Advances and research in the area of Equine Assisted Interventions (Hippotherapy and Therapeutic Riding) have led to a progressive move away from empirical observation to scientific evidence. This is why it is necessary to develop scientific studies that contribute to scientific evidence. This has motivated an international group of experts to design and develop an international clinical trial to collect data on therapeutic horse riding in a group of adults with arthritis. Starting with a pilot project, which is the one presented here.

The established hypothesis is that people diagnosed with arthritis who follow a standardised Therapeutic Riding treatment, as an experimental group, improve their state of health in relation to those who follow a protocolised physical exercise table.

Main objectives: To evaluate the possible changes in the state of health of individuals diagnosed with arthritis who follow a standardised Therapeutic Riding treatment, as an experimental group, versus patients who follow a standardised physical exercise programme and to analyse the effectiveness of the Therapeutic Riding treatment in patients diagnosed with arthritis in terms of pain, joint mobility, static and dynamic balance, gait, capacity for effort and quality of sleep. Furthermore, the aim is to monitor and establish the methodology, protocols and phases in the Therapeutic Riding treatment of patients with a diagnosis of arthritis, as well as to contribute to assessment protocols.

Methodology: In order to achieve the objectives, a double-blind randomised pilot project is proposed in a sample of 10 subjects participating in a therapeutic horse riding programme and 10 subjects participating as a control group in a physical exercise programme. The intervention guidelines for both groups are established in a programme of 12 sessions in total, 6 weeks in duration, twice a week and a duration of 45 minutes each session. All interventions will be carried out by specialist professionals. Pain will be assessed using the EVA scale and questionnaires; joint range in the back, hips, knees and shoulders using goniometry; postural stability using the Romberg test on pressure platforms; gait analysis using inertial sensors during the 10-metre test; capacity for effort using the 2-minute walk test and the use of a smartwatch; and sleep quality using the PittsBurg sleep quality test and MOVOI's TicSleep tool. All assessments are non-invasive.

The project is coordinated by AINISE (International Alliance for Healthy Equine Interaction) and involves an international scientific group led by Dr Íñigo Hernández. It is made up of volunteer expert researchers from 8 countries. Germany, Argentina, Spain, France, Malta, Mexico, Portugal, USA, in which the research group Physioh of the University of Extremadura participates. The project is based on the published trial of Dr. Sharon White Lewis University of Missouri-Kansas City. "A Randomized controlled trial comparing equine-assisted therapy and exercise education for adults and older adults with arthritis". And it is currently supported to start the pilot programme by the Norwegian Ann Kern-Godal Foundation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with arthritis.
* Age over 25 and under 65.
* Not riding on horseback in the last 6 months.
* Enough physical autonomy to be able to ride independently.
* Having pain in a joint with mild to moderate pain and / or decreased range of motion in any joint of a minimum of 10%

Exclusion Criteria:

* Age under 25 and over 65.
* Having ridden on horseback in the previous 6 months.
* NOT having sufficient physical autonomy to be able to ride independently.
* DO NOT have pain in any joint with mild to moderate pain and / or
* DO NOT have a decrease in the range of motion in any joint of a minimum of 10% Have some other associated neuromuscular disease.
* Pregnancy

Contraindications of the E.T.: The German Commissariat for Therapeutic Riding Deutsches Kuratorium Für Therpeutisches Reiten (DKThR) endorse by more than 40 years of research, training and practice of said contraindications in relative and absolute terms, being:

Relative contraindications:

Relative contraindications: It depends on each person. To value. The current relative contraindications always require a detailed consultation with the treating specialist and weighing the risks in Relationship with the expected success of the treatment.

* Hip displacement (the degree must be known).
* Metal implants in the extremities.
* Disc operations (must have passed more than 1 year).
* Degenerative immobilization of the spine (depends on the location).
* Scoliosis Cobb angle> 25º (outside the central straight line).
* M.Bechterew (depends on immobility and pain).
* Osteoporosis (dig with Cortisone and inactivity).
* Hematolytics (Marcumar).
* disturbed blood clotting.
* Spondylolisthesis.
* Epilepsy (the patient would have to spend a year without seizures; you have to think about the type of seizure, the triggering cause, the patient's age and weight).
* Diabetes mellitus (consider age, intensity and coexistence with diabetes). • Rhythmic cardiac disorders.
* Heart failure.
* Heart attack (it must be more than a year since the heart attack).
* Extreme trophic and sensitivity disorders.
* Age (depending on size and evolution, from 4 years to almost 65).
* Obesity (depends on the horses available, and the severity of the limitation of movement).
* Lack of trunk control.
* Seriously disturbed behavior (aggressive patients, with loud voices, etc.). • Periarticular ossifications.
* Bladder catheter.
* Sharp pains.
* Endoprosthesis (knee, hip).

Absolute contraindications:

* Acute inflammatory processes.
* Acute herniated disc prolapse.
* Allergies (dust, horse hair).
* Insurmountable adductor spasticity.
* Coxarthrodesis.
* Acute rheumatism.
* Thrombosis, thrombophlebitis.
* Arterial hypertonia with a tendency to hypertensive crisis.
* Angina pectoris, strong arteriosclerosis.
* Spondylodesis (exception: stable angular spondylodesis in spinal cord injuries, in these usually only one segment stabilizes, talk to the doctor).
* Implants of the trunk, pelvis and femur-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Pain in the main joints including at least back, waist, knees and shoulders | Change from baseline at Week 4 and Week 8
  Analogic visual scale McGill Pain Quetionnaire Functional Pain tests

SECONDARY OUTCOMES:
Joint mobility: back, waist, knees and shoulders | Change from baseline at Week 4 and Week 8
  Joint goniometry. Digital goniometer
Dynamic balance | Change from baseline at Week 4 and Week 8
  Berg balance test
Static balance | Change from baseline at Week 4 and Week 8
  Romberg balance test on pressure platform. To stay standing up during 30 seconds, without moving, eyes open and closed.
Gait | Change from baseline at Week 4 and Week 8
  10 Meters moving test. Assesment by intertial sensors placed in Head, L3, Hip, Tibia and Arms
Exercise capacity | Change from baseline at Week 4 and Week 8
  Two minutes walk test on a 30 meter straight line. Measurement of daily activity with a smartwatch using a heart rate monitor and all watch sensors (subjects will keep watches on their wrist for the entire duration of study)
Sleep quality | Each day from Week 1 at Week 8
  Measurements of the sleeping quality based on the times of the different phases with the tool TicSleep from MOVOI (Smartwatch data collection system)
Sleep quality | Change from baseline at Week 8
  PittsBurg sleeping quality test

CONTACTS AND LOCATIONS:
Overall Officials: Íñigo Hernández Rodríguez, Phd, Study Director — HCU of Vigo
Locations (1):
- María D Apolo Arenas, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo PA, Starling JMP, Oliveira VC, Gontijo APB, Mancini MC. Combining balance-training interventions with other active interventions may enhance effects on postural control in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Braz J Phys Ther. 2020 Jul-Aug;24(4):295-305. doi: 10.1016/j.bjpt.2019.04.005. Epub 2019 May 3. PMID 31076254
- [Background] Caña-Pino, A., Apolo-Arenas, M. D., Moral-Blanco, J., Álvaro-de Diego, J., & Gutiérrez, C. F. (2015). Assessment by accelerometer of postural balance in standing-sitting position in healthy subjects-A pilot study. Fisioterapia, 37(6), 271-278. https://doi.org/10.1016/j.ft.2014.12.004
- [Background] Charry-Sanchez JD, Pradilla I, Talero-Gutierrez C. Animal-assisted therapy in adults: A systematic review. Complement Ther Clin Pract. 2018 Aug;32:169-180. doi: 10.1016/j.ctcp.2018.06.011. Epub 2018 Jun 28. PMID 30057046
- [Background] Fernández-Gutiérrez, C., Apolo-Arenas, M. D., Martínez-García, Y., & Caña-Pino, A. (2015). Effects of hippotherapy on postural stability in cerebral palsy: report of a case. Fisioterapia, 37(3), 135-139.
- [Background] Gutiérrez, C. F., Arenas, M. D. A., Moral-Blanco, J., Madrid-Moreno, M., & Pino, A. C. (2019). Valoración con acelerómetros del incremento en el control postural y equilibrio de una niña con parálisis cerebral que recibe hipoterapia. Cuestiones de fisioterapia: revista universitaria de información e investigación en Fisioterapia, 48(2), 127-132.
- [Background] Hilliere C, Collado-Mateo D, Villafaina S, Duque-Fonseca P, Parraca JA. Benefits of Hippotherapy and Horse Riding Simulation Exercise on Healthy Older Adults: A Systematic Review. PM R. 2018 Oct;10(10):1062-1072. doi: 10.1016/j.pmrj.2018.03.019. Epub 2018 Apr 5. PMID 29626616
- [Background] Mamajón-Pámpano, L., López-Ortiz, L., Pino, A. C., Sánchez-Preciado, A. M., & Arenas, M. D. A. (2019). Study of the effect of sensory dynamic orthosis on postural control in a case of nemaline myopathy. Cuestiones de fisioterapia: revista universitaria de información e investigación en Fisioterapia, 48(3), 228-234.
- [Background] Marquez J, Weerasekara I, Chambers L. Hippotherapy in adults with acquired brain injury: A systematic review. Physiother Theory Pract. 2020 Jul;36(7):779-790. doi: 10.1080/09593985.2018.1494233. Epub 2018 Jul 17. PMID 30015542
- [Background] Massy-Westropp, N. (2004). Measurement of hand joint range of motion in rheumatoid arthritis: Repeatability and variability. Journal of Hand Therapy, 17(4), 438. https://doi.org/10.1197/j.jht.2004.07.027
- [Background] Schmidt J, Wartenberg-Demand A, Forstmeier S. Equine-assisted biographical work (EABW) with individuals in the second half of life: study protocol of a multicentre randomised controlled trial. Trials. 2020 Oct 15;21(1):857. doi: 10.1186/s13063-020-04784-3. PMID 33059730
- [Background] Stergiou A, Tzoufi M, Ntzani E, Varvarousis D, Beris A, Ploumis A. Therapeutic Effects of Horseback Riding Interventions: A Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2017 Oct;96(10):717-725. doi: 10.1097/PHM.0000000000000726. PMID 28252520
- [Background] Tseng SH, Chen HC, Tam KW. Systematic review and meta-analysis of the effect of equine assisted activities and therapies on gross motor outcome in children with cerebral palsy. Disabil Rehabil. 2013 Jan;35(2):89-99. doi: 10.3109/09638288.2012.687033. Epub 2012 May 26. PMID 22630812
- [Background] Villaverde, V., Hernández-García, C., Gonzalez-Alvaro, I., Vargas, E., Abasolo, L., Morado, I. C., & grupo de estudio emAR. (2005). Clinical evaluation of patients with rheumatoid arthritis in Spain. Rev Esp Reumatol, 32(3), 112-120. https://bit.ly/34Tc51z
- [Background] White-Lewis, S. (2018). A Randomized Controlled Trial Comparing Equine-Assisted Therapy and Exercise Education for Adults and Older Adults with Arthritis. Doctoral dissertation, University of Missouri--Kansas City. https://bit.ly/2WOYKE5
- [Background] Zhang L, Cao H, Zhang Q, Fu T, Yin R, Xia Y, Li L, Gu Z. Motion analysis of the wrist joints in Chinese rheumatoid arthritis patients: a cross-sectional study. BMC Musculoskelet Disord. 2018 Jul 28;19(1):270. doi: 10.1186/s12891-018-2146-z. PMID 30055598